CLINICAL TRIAL: NCT05626322
Title: A PHASE 1b/2 STUDY OF PF-07901801, A CD47 BLOCKING AGENT, WITH TAFASITAMAB AND LENALIDOMIDE FOR PARTICIPANTS WITH RELAPSED/REFRACTORY DIFFUSE LARGE B CELL LYMPHOMA NOT ELIGIBLE FOR STEM CELL TRANSPLANTATION
Brief Title: Effects of Maplirpacept (PF-07901801),Tafasitamab, and Lenalidomide in People With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The trial terminated due to the inability to recruit the planned number of subjects. The decision was not based on any safety and/or efficacy concerns
Sponsor: Pfizer (Industry)
Collaborators: MorphoSys AG (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4971003; 2022-502427-21-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL; Lymphoma; Relapsed; Refractory; CD19; CD47; Maplirpacept; Tafasitamab; Lenalidomide
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Recurrence | interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Intervention Model Description: Open label/randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b (Experimental): Participants will be allocated to sequential dose levels of maplirpacept (PF-07901801), administered in combination with standard doses of tafasitamab and lenalidomide, to select two doses for further evaluation in Phase 2. Approximately 20 participants will be enrolled.
  Interventions: Drug: Maplirpacept; Drug: Tafasitamab; Drug: Lenalidomide
- Phase 2 (Experimental): Participants will be randomized to 1 of 2 different dose levels of maplirpacept (PF-07901801) which will be administered in combination with standard doses of tafasitamab and lenalidomide. Approximately 50 participants will be enrolled (25 per dose).
  Interventions: Drug: Maplirpacept; Drug: Tafasitamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Maplirpacept — Intravenous infusion
  Other Names: PF-07901801, TTI-622
Drug: Tafasitamab — Intravenous infusion
  Other Names: Minjuvi, Monjuvi
Drug: Lenalidomide — Oral (by mouth)
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to learn about the effects of three study medicines [maplirpacept (PF-07901801), tafasitamab, and lenalidomide] when given together for the treatment of diffuse large B-cell lymphoma (DLBCL) that:

* is relapsed (has returned after last treatment) or
* is refractory (has not responded to last treatment)

DLBCL is a type of non-Hodgkin lymphoma (NHL). NHL is a cancer of the lymphatic system. It develops when the body makes abnormal lymphocytes. These lymphocytes are a type of white blood cell that normally help to fight infections.

This study is seeking participants who are unable or unwilling to undergo an autologous stem cell transplantation (when doctors put healthy blood cells back into your body) or CAR-T immune cell therapy.

Everyone in this study will receive three medicines: maplirpacept (PF-07901801), tafasitamab and lenalidomide. Participants will receive maplirpacept (PF-07901801) and tafasitamab at the study clinic by intravenous (IV) infusion (given directly into a vein) and lenalidomide will be taken by mouth at home. Study interventions will be administered in 28-day cycles. Maplirpacept (PF-07901801) will be given weekly for the first three cycles and then every two weeks. Tafasitamab will administered on Days 1, 4, 8, 15 and 22 in cycle 1, weekly in cycles 2 and 3 and then every 2 weeks in cycle 4 and beyond. Lenalidomide will be taken every day for Days 1 to 21 of each 28-day cycle for the first 12 cycles.

Participants can continue to take maplirpacept (PF-07901801) and tafasitamab until their lymphoma is no longer responding. Lenalidomide is discontinued after 12 cycles.

Maplirpacept (PF-07901801) will be given at different doses to different participants. Everyone taking part will receive approved doses of tafasitamab and lenalidomide. We will compare the experiences of people receiving different doses of PF-07901801. This will help us to determine what dose is safe and effective when combined with the other 2 study medicines.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 1b/2 study to evaluate the safety, tolerability and potential clinical benefits of maplirpacept (PF-07901801), an anti-CD47 molecule, in combination with standard doses of tafasitamab and lenalidomide in participants with relapsed/refractory (R/R) DLBCL not eligible for or unwilling to undergo high dose chemotherapy and subsequent autologous stem cell transplantation (ASCT) or unable to receive approved chimeric antigen receptor T-cell (CAR-T) therapy (for example, due to logistical limitations).

For Phase 1b, participants must have previously received at least 1 prior systemic treatment regimen. For Phase 2, participants must have received at least 1 but no more than 2 prior systemic treatment regimens. All participants must have previously received an anti-CD20 containing regimen.

Phase 1b will assess dose-limiting toxicities of maplirpacept (PF-07901801) when administered in combination with tafasitamab and lenalidomide, to select up to 2 doses for the Phase 2 part of the study. Phase 2 will evaluate safety and efficacy to determine the recommended Phase 3 dose of Maplirpacept (PF-07901801) to be administered in combination with tafasitamab and lenalidomide.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of DLBCL
* Relapsed or refractory disease
* Participant is not be a candidate for or is unwilling to undergo high dose chemotherapy and subsequent stem cell transplant and/or is unable to receive chimeric antigen receptor (CAR) T-cell therapy
* Previous treatment with at least one prior line of systemic therapy (for phase 2, at least 1 and no more than 2 prior lines of systemic therapy). Prior therapy must include an anti-CD20 antibody.
* Adequate bone marrow, hepatic and renal function
* Eastern Cooperative Oncology Group (ECOG) ≤2
* Must provide a tumor tissue sample (fresh or archival, collected prior to start of treatment) for biomarker analysis

Key Exclusion Criteria:

* Prior treatment with an anti-CD47 or anti-CD19 (other than CAR T) or immunomodulatory agents
* Prior allogeneic stem cell transplantation or autologous stem cell transplantation within 12 weeks prior to enrolment
* Participants with active, uncontrolled bacterial, fungal or viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (4):
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Lifespan Cancer Institute, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
- Yamagata University Hospital, Yamagata, Japan
- South Korea (2):
  - Dong-A University Hospital, Busan, Pusan-kwangyǒkshi
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4971003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 participants were screened of which 3 participants failed screening, and 6 participants were enrolled and received study treatment.
Pre-assignment Details: The study was planned to be conducted in 2 parts: phase 1b dose escalation and phase 2 dose expansion. Phase 2 of the study was not initiated per business decision made by Sponsor; hence, data for Phase 2 is not reported in any part of the record.
Groups:
- PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide: Participants with relapsed/refractory diffuse large B cell lymphoma received PF-07901801 4 milligrams per kilogram (mg/kg) as an intravenous (IV) infusion once weekly (QW) during Cycle 1 to 3 followed by twice weekly (Q2W) dosing from Cycle 4 onwards along with tafasitamab 12 mg/kg as an IV infusion on Days 1, 4, 8, 15 and 22 of Cycle 1, QW during Cycle 2 and 3 and Q2W from Cycle 4 onwards. Participants were administered lenalidomide 25 milligrams (mg) by mouth (PO) on Days 1 through 21 of each cycle for up to 12 cycles. Each Cycle = 28 Days. Participants received treatment until disease progression, start of new anti-cancer therapy or death, whichever occurred first.
- PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide: Participants with relapsed/refractory diffuse large B cell lymphoma received PF-07901801 10 mg/kg as an IV infusion QW during Cycle 1 to 3 followed by Q2W dosing from Cycle 4 onwards along with tafasitamab 12 mg/kg as an IV infusion on Days 1, 4, 8, 15 and 22 of Cycle 1, QW during Cycle 2 and 3 and Q2W from Cycle 4 onwards. Participants were administered lenalidomide 25 mg PO on Days 1 through 21 of each cycle for up to 12 cycles. Each Cycle = 28 Days. Participants received treatment until disease progression, start of new anti-cancer therapy or death, whichever occurred first.
- PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide: Participants with relapsed/refractory diffuse large B cell lymphoma received PF-07901801 18 mg/kg as an IV infusion QW during Cycle 1 to 3 followed by Q2W dosing from Cycle 4 onwards along with tafasitamab 12 mg/kg as an IV infusion on Days 1, 4, 8, 15 and 22 of Cycle 1, QW during Cycle 2 and 3 and Q2W from Cycle 4 onwards. Participants were administered lenalidomide 25 mg PO on Days 1 through 21 of each cycle for up to 12 cycles. Each Cycle = 28 Days. Participants received treatment until disease progression, start of new anti-cancer therapy or death, whichever occurred first.
Period: Overall Study
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Started | 3 | 2 | 1
Completed | 0 | 0 | 0
Not Completed | 3 | 2 | 1
Not completed — Death | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Progressive Disease | 0 | 1 | 1
Not completed — Study terminated by sponsor | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide: Participants with relapsed/refractory diffuse large B cell lymphoma received PF-07901801 4 mg/kg as an IV infusion QW during Cycle 1 to 3 followed by Q2W dosing from Cycle 4 onwards along with tafasitamab 12 mg/kg as an IV infusion on Days 1, 4, 8, 15 and 22 of Cycle 1, QW during Cycle 2 and 3 and Q2W from Cycle 4 onwards. Participants were administered lenalidomide 25 mg PO on Days 1 through 21 of each cycle for up to 12 cycles. Each Cycle = 28 Days. Participants received treatment until disease progression, start of new anti-cancer therapy or death, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide | Total
Number analyzed (Participants) | 3 | 2 | 1 | 6
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-44 years | 0 | 0 | 1 | 1
  Age: 45-64 years | 1 | 2 | 0 | 3
  Age: >=65 years | 2 | 0 | 0 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants] — Data for arm - ''PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide'' is not disclosed to avoid risk of identification and kept under ''Not disclosed'' category.
  Participants
    Gender: Female | 2 | 0 | 0 | 2
    Gender: Male | 1 | 2 | 0 | 3
    Gender: Not disclosed | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data for arm - ''PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide'' is not disclosed to avoid risk of identification and kept under ''Not disclosed'' category.
  Participants
    Race: White | 1 | 2 | 0 | 3
    Race: Black or African American | 1 | 0 | 0 | 1
    Race: Asian | 1 | 0 | 0 | 1
    Race: Not disclosed | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data for arm - ''PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide'' is not disclosed to avoid risk of identification and kept under ''Not disclosed'' category.
  Participants
    Ethnicity: Not Hispanic or Latino | 3 | 2 | 0 | 5
    Ethnicity: Not disclosed | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs included: Hematological: Grade (G) 4 thrombocytopenia (<25,000/microliter [mcL]) lasting >=72 hours or a platelet count <=10,000/mcL at any time, unexplained by underlying disease; >=G3 thrombocytopenia associated with >=G2 bleeding, unexplained by underlying disease. G4 anemia; unexplained by underlying disease; G4 neutropenia lasting >=7 days, unexplained by underlying disease; G3 febrile (>38.3-degree Celsius [C]) neutropenia lasting >=7 days, unexplained by underlying disease; G4 febrile neutropenia unexplained by underlying disease. Non-hematological: any treatment-related >=G3 non-hematologic toxicity; Other >=G2 PF-07901801-related non-hematologic toxicities that, in the opinion of the investigator, required a dose reduction or discontinuation of PF-07901801 were considered a DLT.
Time Frame: Cycle 1 (28 Days)
Population: DLT evaluable set included all enrolled participants who received at least 1 dose of the study treatment in the Phase 1b of the study and either experienced DLTs or completed the DLT observation period without DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 2 | 2 | 1
Participants | 0 | 0 | 0

2. Secondary Outcome: Phase 1b: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs are those events with onset dates occurred during the on-treatment period for the first time, or if the worsening of an event is during the on-treatment period.
Time Frame: From Day 1 of dosing up to 35 days post last dose of PF-07901801 and/or lenalidomide or 90 days after the last dose of tafasitamab, whichever was longer (maximum up to 14.2 months of exposure)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 1
Participants | 3 | 2 | 1

3. Secondary Outcome: Phase 1b: Number of Participants With Serious Treatment Emergent Adverse Events
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/ incapacity, was a congenital anomaly/birth defect or other important medical event. TEAEs are those events with onset dates occurred during the on-treatment period for the first time, or if the worsening of an event is during the on-treatment period.
Time Frame: as for outcome 2
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 1
Participants | 3 | 0 | 0

4. Secondary Outcome: Phase 1b: Number of Participants With Treatment-Related AEs
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Related AEs were those related to any study drug (i.e., at least one of the study drugs) reported by the investigator.
Time Frame: as for outcome 2
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 1
Participants | 3 | 2 | 1

5. Secondary Outcome: Phase 1b: Number of Participants With Grade Shift From Baseline in Hematology Parameters to Any Time Post-baseline
Description: The following hematological parameters were assessed: anemia, hemoglobin increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, and white blood cell (WBC) decreased. Lab abnormalities were graded according to National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) version (v) 5.0 where Grade 0= no AE, Grade 1= mild AE, Grade 2 =moderate AE, Grade 3= severe AE, and Grade 4= life-threatening consequences; urgent intervention indicated. Only those parameters with at least 1 non-zero data values showing any shift in grades from Baseline to any time post-baseline in any reporting group were reported in this outcome measure. Participants whose grade category was unchanged (e.g. Grade 0 to Grade 0) were not reported.
Time Frame: From baseline (latest non-missing value from pre-treatment period) up to 35 days post last dose of PF-07901801 and/or lenalidomide or 90 days after the last dose of tafasitamab, whichever was longer (maximum up to 14.2 months of exposure)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 1
Participants
  Anemia: Grade 1 to Grade 2 | 1 | 0 | 0
  Anemia: Grade 2 to Grade 3 | 1 | 0 | 0
  Leukocytosis: Grade 0 Grade 3 | 1 | 0 | 0
  Lymphocyte count decreased: Grade 0 to Grade 2 | 0 | 1 | 1
  Lymphocyte count decreased: Grade 0 to Grade 3 | 1 | 0 | 0
  Lymphocyte count decreased: Grade 1 to Grade 2 | 1 | 0 | 0
  Lymphocyte count decreased: Grade 1 to Grade 3 | 0 | 1 | 0
  Lymphocyte count increased: Grade 0 Grade 2 | 1 | 0 | 0
  Neutrophil count decreased: Grade 0 to Grade 2 | 0 | 1 | 1
  Neutrophil count decreased: Grade 0 to Grade 3 | 2 | 1 | 0
  Neutrophil count decreased: Grade 0 to Grade 4 | 1 | 0 | 0
  Platelet count decreased: Grade 0 to Grade 1 | 2 | 0 | 1
  Platelet count decreased: Grade 0 to Grade 4 | 0 | 1 | 0
  Platelet count decreased: Grade 1 to Grade 4 | 1 | 0 | 0
  WBC decreased: Grade 0 to Grade 1 | 0 | 1 | 1
  WBC decreased: Grade 0 to Grade 2 | 0 | 1 | 0
  WBC decreased: Grade 0 to Grade 4 | 1 | 0 | 0
  WBC decreased: Grade 1 to Grade 2 | 1 | 0 | 0

6. Secondary Outcome: Phase 1b: Number of Participants With Grade Shift From Baseline in Chemistry Parameters to Any Time Post Baseline
Description: The following clinical chemistry parameters were assessed: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatinine increased, hypercalcemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia and hyponatremia. Lab abnormalities were graded according to NCI CTCAE v5.0 where Grade 0= no AE, Grade 1=mild AE, Grade 2 = moderate AE, Grade 3 =severe AE, and Grade 4 =life-threatening consequences; urgent intervention indicated. Only those parameters with at least 1 non-zero data values showing any shift in grades from Baseline to any time post-baseline in any reporting group were reported in this outcome measure. Participants whose grade category was unchanged (e.g. Grade 0 to Grade 0) were not reported.
Time Frame: as for outcome 5
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 1
Participants
  Alanine aminotransferase increased: Grade 0 to Grade 1 | 1 | 1 | 1
  Alanine aminotransferase increased: Grade 1 to Grade 0 | 0 | 1 | 0
  Alkaline phosphatase increased: Grade 0 to Grade 1 | 2 | 1 | 0
  Alkaline phosphatase increased: Grade 1 to Grade 0 | 1 | 0 | 0
  Aspartate aminotransferase increased: Grade 0 to Grade 1 | 1 | 2 | 0
  Blood bilirubin increased: Grade 0 to Grade 1 | 1 | 0 | 0
  Blood bilirubin increased: Grade 0 to Grade 2 | 1 | 0 | 0
  Creatinine increased: Grade 0 to Grade 1 | 0 | 1 | 0
  Creatinine increased: Grade 0 to Grade 3 | 1 | 0 | 0
  Creatinine increased: Grade 1 to Grade 2 | 1 | 0 | 0
  Hypercalcemia: Grade 0 to Grade 1 | 1 | 0 | 0
  Hyperkalemia: Grade 0 to Grade 1 | 1 | 0 | 0
  Hypermagnesemia: Grade 0 to Grade 1 | 0 | 1 | 0
  Hypernatremia: Grade 0 to Grade 1 | 1 | 0 | 0
  Hypoalbuminemia: Grade 1 to Grade 2 | 1 | 0 | 0
  Hypoalbuminemia: Grade 1 to Grade 3 | 1 | 0 | 0
  Hypocalcemia: Grade 0 to Grade 1 | 2 | 1 | 0
  Hypokalemia: Grade 0 to Grade 2 | 3 | 0 | 0
  Hypomagnesemia: Grade 0 to Grade 1 | 1 | 0 | 0
  Hypomagnesemia: Grade 0 to Grade 2 | 1 | 0 | 0
  Hyponatremia: : Grade 0 to Grade 1 | 3 | 0 | 0

7. Secondary Outcome: Phase 1b: Percentage of Participants With Objective Response (OR) as Per Lugano Response Classification Criteria 2014 as Assessed by the Investigator
Description: OR:best overall response (BOR) of complete response (CR) or partial response (PR) per Lugano Response Classification Criteria 2014 as determined by investigator. CR:positron emission tomography-computed tomography (PET-CT) score 1 (complete metabolic response), 2 (likely benign), or 3 (uncertain significance) with or without a residual mass on Deauville five-point scale ([5PS] standardized scoring system used to evaluate the extent of disease activity in patients with lymphoma through PET scans, ranging from 1 to 5, higher scores indicates more disease activity) or on computed tomography (CT),target nodes/nodal masses regressed to <=1.5 centimeter (cm) in longest diameter (LDi). PR:PET-CT score 4 (possible residual disease) or 5 (progressive disease) with reduced uptake compared with baseline and residual mass(es) of any size or On CT >=50% decrease in sum of the product of the diameters (SPD) of up to 6 target measurable nodes and extra nodal sites. 95% CI was based on Wilson method.
Time Frame: From date of first dose until first documentation of disease progression (PD), death or start of new anticancer therapy, whichever occurred first (maximum up to 14.2 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 1
Percentage of participants | 66.7 [12.5 to 98.2] | 100.0 [19.8 to 100.0] | 0 [0 to 94.5]

8. Secondary Outcome: Phase 1b: Duration of Response (DoR) as Per Lugano Response Classification Criteria 2014 as Assessed by the Investigator
Description: DoR: time from first documentation of OR until PD, or death due to any cause, whichever occurred first. DoR was censored on date of last adequate disease assessment for participants without an event. OR=BOR of CR or PR,CR=PET-CT score 1,2,or 3 with/without a residual mass on Deauville five-point scale(1 to 5,higher scores=more disease activity)or on CT,target nodes/nodal masses regressed to <=1.5cm in LDi. PR:PET-CT score 4 or 5 with reduced uptake compared with baseline and residual mass of any size or On CT >=50% decrease in SPD of up to 6 target measurable nodes and extra nodal sites. PD:PET-CT score 4 or 5 with increase in intensity of uptake from baseline and/or new fluorodeoxyglucose (FDG)-avid foci consistent with lymphoma at interim or end-of-treatment assessment or on CT,an individual abnormal node/lesion with: LDi>1.5cm and increase by >=50% from product of perpendicular diameters nadir and increase in LDi or SDi from nadir 0.5cm for lesions <=2cm and 1.0cm for lesions >2cm.
Time Frame: From first documentation of OR until PD or death due to any cause whichever occurred first or date of censoring (maximum up to 14.2 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Only participants with objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 2 | 2 | 0
Months | 11.9 [9.6 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [3.3 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. |

9. Secondary Outcome: Phase 1b: Percentage of Participants With CR as Per Lugano Response Classification Criteria 2014 as Assessed by the Investigator
Description: CR as per Lugano Response Classification Criteria 2014 as assessed by the investigator was defined as: PET-CT score 1 (complete metabolic response), 2 (likely benign), or 3 (uncertain significance) with or without a residual mass on 5PS (standardized scoring system used to evaluate the extent of disease activity in patients with lymphoma through PET scans, ranging from 1 to 5, higher scores indicates more disease activity) or on CT, target nodes/nodal masses regressed to <=1.5 cm in LDi.
Time Frame: From date of first dose until first documentation of CR (maximum up to 14.2 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 1
Percentage of participants | 66.7 [12.5 to 98.2] | 100.0 [19.8 to 100.0] | 0.0 [NA to NA] — Upper and lower limit of 95% CI could not be estimated due to insufficient number of participants with events.

10. Secondary Outcome: Phase 1b: Duration of Complete Response (DoCR) as Per Lugano Response Classification Criteria 2014 as Assessed by the Investigator
Description: DoCR:time from first documentation of CR until PD,or death, whichever occurred first. CR:PET-CT 1(complete metabolic response),2(likely benign),3(uncertain significance)with or without residual mass on 5PS(scale from 1 to 5,higher scores=more disease activity)/CT,target nodes/nodal masses regressed <=1.5cm in LDi.PD:PET-CT 4(possible residual disease)or 5(PD)with increase intensity of uptake and new FDG-avid foci consistent with lymphoma at interim/EOT assessment/CT,individual abnormal node/lesion with:LDi >1.5cm and increase >=50% from PPD nadir, increase in LDi or SDi from nadir 0.5cm for lesions <=2cm and 1.0cm for lesions >2cm. DoCR censored on date of last adequate assessment for participants without an event on date of last adequate disease assessment before new anti-cancer therapy if new anti-cancer therapy started prior to event,date of last adequate disease assessment before 2 or more missing disease assessments for participants with event after 2 or more missing assessments.
Time Frame: From time of first documentation of CR until PD, or death due to any cause, whichever occurred first or date of censoring (maximum up to 14.2 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Only participants with complete response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 2 | 2 | 0
Months | 11.9 [9.6 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [3.3 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. |

11. Secondary Outcome: Phase 1b: Progression Free Survival (PFS) as Per Lugano Response Classification Criteria 2014 as Assessed by the Investigator
Description: PFS: time from date of first dose until PD per Lugano Response Classification Criteria 2014 or death due to any cause,whichever occurred first.Participants without any event,censored on date of last adequate disease assessment;participants with new anticancer therapy prior to an event,censored on date of last disease assessment before new anticancer therapy;participants with an event after a gap of 2 or more missing disease assessments,censored on date of last disease assessment before gap;participants without an adequate post-baseline disease assessment were censored on date of first dose of study intervention unless death occurred on or before time of second planned disease assessment in which case death was considered an event.PD:PET-CT score 4 or 5 with increase in intensity of uptake from baseline and/or new FDG or LDi>1.5cm and increase by >=50% from product of perpendicular diameters nadir and increase in LDi or SDi from nadir 0.5cm for lesions <=2cm and 1.0cm for lesions >2cm.
Time Frame: From date of first dose until PD or death due to any cause, whichever occurred first or censoring date (maximum up to 14.2 months)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 1
Months | 13.7 [11.4 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | NA [5.6 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient number of participants with events. | 1.2 [NA to NA] — Upper and lower limit of 95% CI could not be estimated due to insufficient number of participants with events.

12. Secondary Outcome: Phase 1b: Plasma Concentration of PF-07901801
Description: All concentrations assayed below the level of quantification (BLQ) were set to 0 and their data is not reported in this outcome measure.
Time Frame: Cycle 1 and 2 Day 1: Predose, 1 Hour (H) and 5H post dose; Cycle 1 Day 8: pre-dose, Day 1 of Cycles 3, 4, 5, 7, 10 and 13: Predose
Population: The Pharmacokinetic (PK) analysis set included all participants in the safety analysis set who had at least 1 post-dose concentration measurement. Here, "Number Analyzed" signifies number of participants evaluable at specified timepoints. The participant in PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide withdrew consent hence, the "Overall Number of Participants Analyzed" is reported as 0.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 0
Micrograms per milliliter
  Cycle 1 Day 1: Predose: number analyzed (Participants) | 0 | 1 | 0
  Cycle 1 Day 1: Predose |  | 0.1 (NA) — Geometric coefficient of variation was not estimated as only 1 participant was analyzed. |
  Cycle 1 Day 1: 1 hour | 64.3 (45) | 213.4 (31) |
  Cycle 1 Day 1: 5 hours | 50.7 (47) | 194.2 (42) |
  Cycle 1 Day 8: Predose | 4.0 (159) | 21.1 (85) |
  Cycle 2 Day 1: Predose | 7.9 (201) | 88.3 (35) |
  Cycle 2 Day 1: 1 hour | 75.3 (63) | 308.1 (42) |
  Cycle 2 Day 1: 5 hours | 67.6 (71) | 276.4 (31) |
  Cycle 3 Day 1: Predose | 10.9 (168) | 130.4 (10) |
  Cycle 4 Day 1: Predose | 15.0 (190) | 75.1 (110) |
  Cycle 5 Day 1: Predose | 2.0 (57) | 35.2 (187) |
  Cycle 7 Day 1: Predose: number analyzed (Participants) | 2 | 2 | 0
  Cycle 7 Day 1: Predose | 2.3 (20) | 21.0 (50) |
  Cycle 10 Day 1: Predose: number analyzed (Participants) | 2 | 1 | 0
  Cycle 10 Day 1: Predose | 2.0 (15) | 28.6 (NA) — Geometric coefficient of variation was not estimated as only 1 participant was analyzed. |
  Cycle 13 Day 1: Predose: number analyzed (Participants) | 2 | 1 | 0
  Cycle 13 Day 1: Predose | 1.6 (83) | 26.9 (NA) — Geometric coefficient of variation was not estimated as only 1 participant was analyzed. |

13. Secondary Outcome: Phase 1b: Number of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibodies (NAb) Against PF-07901801
Description: Number of participants with ADA and NAb against PF-07901801 were reported in this outcome measure. A participant was ADA (or NAb) positive if: (1) baseline titer was missing or negative and participant had >= 1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a >= 4-folder dilution increase in titer from baseline in >= 1 post-treatment sample (treatment-boosted).
Time Frame: From first dose of the study treatment (Day 1) up to end of study treatment (maximum up to 14.2 months)
Population: Immunogenicity analysis set included all participants in the safety analysis set who had at least 1 sample tested for ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
Number analyzed (Participants) | 3 | 2 | 1
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 of dosing up to 35 days post last dose of PF-07901801 and/or lenalidomide or 90 days after the last dose of tafasitamab, whichever was longer (maximum up to 14.2 months of exposure)
Description: Same event may appear as non-SAE and SAE, however, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all enrolled participants who received at least 1 dose of study treatment.
Arm/Group | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide
All-Cause Mortality (participants affected / at risk) | 2/3 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/3 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide (N=3) | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide (N=2) | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide (N=1)
Appendicitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-07901801 4 mg/kg + Tafasitamab + Lenalidomide (N=3) | PF-07901801 10 mg/kg + Tafasitamab + Lenalidomide (N=2) | PF-07901801 18 mg/kg + Tafasitamab + Lenalidomide (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gingival ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Oral infection (Infections and infestations) | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 1 | 0
Platelet count decreased (Investigations) | 2 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 2 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor (or its agents) has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT05626322/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT05626322/SAP_001.pdf